CLINICAL TRIAL: NCT04529577
Title: His-bundle Pacing vs. Right Ventricular Apical Pacing in Patients With Reduced Ejection
Brief Title: His-bundle Pacing vs. Right Ventricular Apical Pacing in Patients With Reduced Ejection Fraction
Acronym: HIS-PrEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HIS-PrEF_study
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-02

CONDITIONS: His Bundle Pacing; Heart Failure, Systolic
Keywords: His bundle pacing; Conduction system pacing; Heart failure, systolic; Quality of life; Left ventricular ejection fraction
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Intervention Model Description: Randomized double blinded crossover design.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients and outcomes assessors are blinded. Staff involved in device programming are not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- His-bundle pacing first (Experimental): Patients are allocated to receive His-bundle pacing for a period of 6 months. Then the patients will cross over to traditional right ventricular (RV) apical pacing for 6 months.
  Interventions: Device: His-bundle pacing
- RV apical pacing first (Experimental): Patients are allocated to receive traditional RV apical pacing for a period of 6 months. Then the patients will cross over to His-bundle pacing for 6 months.
  Interventions: Device: His-bundle pacing

INTERVENTIONS:
Device: His-bundle pacing — A standard pacing electrode (Medtronic 4076) will be placed in RV apex (or RV septum as a secondary option) and in the right atrial appendage (if indicated).
  A dedicated His-bundle pacemaker electrode (Medtronic 3830) will be placed in the region of His bundle, using a dedicated introducer sheath (Medtronic C304 or Medtronic C315). His-bundle potentials will be identified and His-bundle capture (non-selective or selective) will be ascertained using an electrophysiology recording system. Device programming will focus on providing physiological atrioventricular delay and safety RV pacing as backup.

SUMMARY:
The study compares standard right ventricle apical pacing with so called His-bundle pacing, for patients with slightly or moderately reduced ejection fraction and atrioventricular block requiring pacemaker therapy. The primary outcome is left ventricular ejection fraction measured after 6 months.

DETAILED DESCRIPTION:
Patients with reduced systolic ejection fraction (40≤ ejection fraction ≤55%) and pacemaker indication due to high degree AV block are included. The study has a randomized double blinded crossover design. Patients are implanted with a standard right ventricle lead and right atrial lead (if indicated), and in addition a His-bundle lead. Randomization is performed as to which pacing modality is used during the first 6 months. After 6 months the pacing modality is changed. Patients are blinded and endpoint adjudicators, including echocardiography staff, are blinded. Device nurse and physician are not blinded.

Primary endpoint is difference in left ventricular ejection fraction after 6 months, paired comparisons are used and each patient is their own control. Secondary endpoints include complications and safety of the device/electrode, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* AV block II or III with high expected pacing need
* Left ventricular ejection fraction between 40% and 55% (inclusive)
* Willing to participate and sign informed consent

Exclusion Criteria:

* Under 18 years old
* Pregnant
* Hypertrophic cardiomyopathy
* Cardiac sarcoidosis
* Cardiac amyloidosis
* Previous myocardial infarction within last 3 months
* Ventricular septum defect or other other left ventricular corrective surgery
* Congenital heart disease surgically corrected
* Atrial fibrillation with uncontrolled rate (if not planned for AV node ablation)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Ejection Fraction | 6 months
  Absolute difference in left ventricular systolic ejection fraction (absolute percent)

SECONDARY OUTCOMES:
Adverse events | 12 months
  Percentage of device-related adverse events. Events will be classified as general, associated with His-bundle lead or associated with RV lead
Left ventricular activation time | 6 months
  Total left ventricular mechanical activation time (measured with tissue doppler echocardiography)
NT-ProBNP | 6 months
  Difference in NT-ProBNP levels
QRS duration | 6 months
  Difference in total QRS duration on ECG
Left Ventricular Activation Time (LVAT) | 6 months
  Maximum unipolar spike-to-peak-T-wave in V5-V6
6 minute walk test | 6 months
  Difference in six minute hall walk test (meters)
Change in quality of life measured by the Short Form Health Survey (SF-36) mean score | 6 months
  Difference in health related quality of life, measured by the SF-36 questionnaire, calculated as difference in mean from baseline to follow-up (calculated using the official scoring algorithm, where each sub scale is assigned a score between 0-100, higher score represents better health)
Change in quality of life measured by the EuroQol EQ-5D-5L Questionnaire | 6 months
  Difference in health related quality of life, measured by the mean score of the EQ-5D (version 5L) questionnaire (totalt score ranging from 5-25 points, higher score represents more health related problems/disability)

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Borgquist, MD PhD, Principal Investigator — Lund University, Skane University Hospital, Arrhythmia Section, Lund, Sweden
Locations (3):
- Sweden (3):
  - Skane University Hospital, Lund
  - Norrland University Hospital, Umeå
  - Region Hallands Sjukhus Varberg, Varberg

IPD SHARING:
Plan to Share IPD: No